CLINICAL TRIAL: NCT03887507
Title: The Implementation of a Reflex Locomotion Program According to Vojta Produces Short-term Automatic Postural Control Changes in Patients With Multiple Sclerosis.
Brief Title: Vojta Therapy in Multiple Sclerosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NUMEN Foundation (Other)
Collaborators: Multiple Sclerosis Foundation of Madrid (Unknown); Fisiovillalba Clinical center (Unknown)
Responsible Party: Principal Investigator, Luis Perales Lopez, Physiotherapy service coordinator, NUMEN Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUMEN
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis; Physical Therapy
Keywords: Vojta therapy; core stability; postural balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): There will be 3 Vojta therapy sessions conducted on 2 consecutive weeks with an interval of 7 dayssessions, on 1st, 7th and 14th days. Each session will consist of a 45-minute Vojta thera between py protocol based on three exercises, 15 minutes per exercise: Crawling Réflex, and 1st phase and 2nd phase Rolling reflex. The relative or close person will be instructed to carry out an exercise protocol to do at home every day for 20 minutes during the 2-week study. All interventions will be made by the principal investigator.
  Interventions: Other: Vojta Therapy
- Standard Therapy (Active Comparator): The standard group shall perform 4 sessions of physiotherapy in the same period for two consecutive weeks, with one hour per session in its specialized MS association, on 1st, 3rd, 8th, 10th and 15th days. This will be applied by experienced physiotherapists during the treatment of people with MS. The program will consist in balance exercises targeting core stability, exercises of coordination and Pilates as well as individual sessions using the Bobath concept. Patients in this group will walk at least for 20 minutes per day during the study period.
  Interventions: Other: Standard Program

INTERVENTIONS:
Other: Vojta Therapy — Each session will consist of a 45-minute Vojta thera between py protocol based on three exercises, 15 minutes per exercise: Crawling reflex, and 1st phase and 2nd phase Rolling reflex.
  Arms: Experimental
Other: Standard Program — The program consist in balance exercises targeting core stability, exercises of coordination and Pilates as well as individual sessions using the Bobath concept.
  Arms: Standard Therapy

SUMMARY:
This Study evaluates the effectiveness of a Vojta locomotion reflex program as short-term automatic postural control in patients with Multiple sclerosis

DETAILED DESCRIPTION:
In two consecutive weeks two interventions will be conducted: Vojta group(A) and standard therapy group(B). The last one is based on balance exercises targeting core stability, Bobath concept and sensory strategies. In the Vojta group 5 sessions will be conducted for a duration of 2 weeks and the same will be realised on the standard group. In addition, during the study, a daily activity shall be prescribed in both groups: Vojta exercise during 20 minutes for group A and walking for 20 minutes in group B.

ELIGIBILITY:
Inclusion Criteria:

* Final diagnosis of MS according to McDonald criteria.
* Walkability with or without assistance (4.0 to 6.5 in EDSS) and dysfunctions defined by the inability to hold the tandem position for 30 seconds with the arms close to body.
* Older than 18 years-old.
* Escorted sessions, a family member or close person.

Exclusion Criteria:

* Phase outbreak or outbreak in the 3 months before the study.
* Medication that prevents or limits the performance of the Locomotion reflex.
* Participation in other studies during the conduct of this study.
* Score inferior to 6 in the Abbreviated Mental Test that prevents understanding of the study consent or that limits the understanding of the test during its realisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 2 weeks
  This test measures the automatic postural control. The Berg scale comprises 14 items (score included 0-4). The total scores can range from 0 (severely affected balance) to 56 (excellent balance).
10 metres walk | 2 weeks
  This Test measures the speed during 10 meter walking at normal pace

SECONDARY OUTCOMES:
Tandem 6 metres test | 2 weeks
  This test measures the balance when walking with one foot in front of the other

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Valdez Palmero, Degree, Study Chair — Rehabilitation Clinic Fisiovillalba; Laura Garcia Ruano, coordinator, Study Chair — Multiple Sclerosis Foundation of Madrid
Locations (1):
- NUMEN Foundation, Madrid, España, Spain

REFERENCES:
- [Derived] Lopez LP, Palmero NV, Ruano LG, San Leon Pascual C, Orile PW, Down AV, Gor Garcia-Fogeda MD, Tore S. The implementation of a reflex locomotion program according to Vojta produces short-term automatic postural control changes in patients with multiple sclerosis. J Bodyw Mov Ther. 2021 Apr;26:401-405. doi: 10.1016/j.jbmt.2021.01.001. Epub 2021 Jan 9. PMID 33992274